CLINICAL TRIAL: NCT05888649
Title: Community Preparedness for Outbreak Response and Readiness for ZEBOV Vaccination in Liberia
Brief Title: Community Preparedness for Outbreak Response and Readiness for Ebola Vaccination in Liberia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: UL-PIRE Africa Center (Other)
Collaborators: West African Consortium for Clinical Research on Epidemic Pathogens (WAC-CREP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: MISP 101054
Record Dates: First submitted 2023-04-27; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Ebola Virus Disease
Keywords: Community Preparedness; Outbreak Response; Ebola Virus Disease (EVD); Ebola Vaccine; Ebola Vaccine Acceptance; Community Leaders; Liberia
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cluster 1: Communities highly affected and impacted by EVD
  Interventions: Behavioral: Community Clusters
- Cluster 2: Communities not highly affected and impacted by EVD
  Interventions: Behavioral: Community Clusters
- Cluster 3: Communities receptive to EVD vaccination
  Interventions: Behavioral: Community Clusters
- Cluster 4: Communities resistance to EVD vaccination
  Interventions: Behavioral: Community Clusters

INTERVENTIONS:
Behavioral: Community Clusters — Assessment of the determinants for community preparedness to EVD outbreaks and acceptance of EVD vaccines.
  Other Names: Community Cohorts

SUMMARY:
This community-based mixed methods study intends to identify, explore, and assess the determinants of community preparedness for outbreak situations, including acceptance for Ebola vaccines.

DETAILED DESCRIPTION:
This community-based study intends to identify, explore, and assess the determinants of community preparedness for outbreak situations and acceptance for the administration of Ebola vaccination. The investigators will conduct an anthropologically driven mixed methods study design that comprises both qualitative and quantitative research methods for the successful implementation of this community-based study. The investigators will conduct structured interviews with community members and local responders to broadly assess and understand the perspectives regarding appropriate strategies previously employed to effectively support community preparedness during outbreak response and also to broadly access and understand appropriate strategies previously employed to effectively support community acceptance for Ebola vaccines, respectively. Learning from the experiences of local voices produces globally emergent systems that are trusted, reliable and sustainable.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Community Leaders
* Community Members
* Reside in 1 of 3 highly prevalent counties
* Participated actively in EVD outbreaks related activities
* Documented roles recognized by the Incident Management System

Exclusion Criteria:

* Not Adults
* Does not reside in any of the 3 highly prevalent counties
* Did not actively participate in the EVD outbreak response related activities
* Roles not documented by the Incident Management System

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health adults (males and females)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Measure #1 | 2 Years
  Assess Community Preparedness with the Resiliency Scale
Measure #2 | 2 Years
  Assess Community Acceptance of EVD Vaccine with the Resiliency Scale

SECONDARY OUTCOMES:
Measure #3 | 2 Years
  Assess Roles of Community Leaders with the Resiliency Scale
Measure #4 | 2 Years
  Assess Roles of Formal and Informal Community Structures with the Resiliency Scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Kennedy, MD, MPH, Principal Investigator — UL-PIRE Africa Center, University of Liberia
Locations (1):
- Montserrado, Margibi and Lofa Counties, Monrovia, Montserrado County, Liberia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kennedy SB, Neaton JD, Lane HC, Kieh MW, Massaquoi MB, Touchette NA, Nason MC, Follmann DA, Boley FK, Johnson MP, Larson G, Kateh FN, Nyenswah TG. Implementation of an Ebola virus disease vaccine clinical trial during the Ebola epidemic in Liberia: Design, procedures, and challenges. Clin Trials. 2016 Feb;13(1):49-56. doi: 10.1177/1740774515621037. Epub 2016 Jan 14. PMID 26768572
- [Result] Nyenswah T, Fallah M, Sieh S, Kollie K, Badio M, Gray A, Dilah P, Shannon M, Duwor S, Ihekweazu C, Cordier-Lassalle T, Shinde SA, Hamblion E, Davies-Wayne G, Ratnesh M, Dye C, Yoder JS, McElroy P, Hoots B, Christie A, Vertefeuille J, Olsen SJ, Laney AS, Neal JJ, Yaemsiri S, Navin TR, Coulter S, Pordell P, Lo T, Kinkade C, Mahoney F; Centers for Disease Control and Prevention (CDC). Controlling the last known cluster of Ebola virus disease - Liberia, January-February 2015. MMWR Morb Mortal Wkly Rep. 2015 May 15;64(18):500-4. PMID 25974635
- [Result] O'Dowd A. Infectious diseases are spreading more rapidly than ever before, WHO warns. BMJ. 2007 Sep 1;335(7617):418. doi: 10.1136/bmj.39318.516968.DB. No abstract available. PMID 17762021
- [Result] Kennedy SB, Nisbett RA. The Ebola epidemic: a transformative moment for global health. Bull World Health Organ. 2015 Jan 1;93(1):2. doi: 10.2471/BLT.14.151068. No abstract available. PMID 25558097
- [Result] Fregonese F. Community involvement in biomedical research conducted in the global health context; what can be done to make it really matter? BMC Med Ethics. 2018 Jun 15;19(Suppl 1):44. doi: 10.1186/s12910-018-0283-4. PMID 29945597
- [Result] Dickert N, Sugarman J. Ethical goals of community consultation in research. Am J Public Health. 2005 Jul;95(7):1123-7. doi: 10.2105/AJPH.2004.058933. Epub 2005 Jun 16. PMID 15983268
- [Result] Wills C, Tyeku V. Community participation is essential in clinical trials. BMJ. 2000 Sep 30;321(7264):833. No abstract available. PMID 11009541
- [Result] Esangbedo DO, Ughasoro MD, Tagbo BN, Olowu A, Anikene C, Iwegbulam CC. Health-Care Workers' Perspectives on Ebola Virus Vaccine: A Focus Group and In-Depth Interview Interventional Study. Am J Trop Med Hyg. 2016 Sep 7;95(3):654-62. doi: 10.4269/ajtmh.16-0206. Epub 2016 Jul 5. PMID 27382077
- [Result] Chiam AL, Cheng NWI, Larson H. Community engagement for outbreak preparedness and response in high-income settings: A systematic review. Glob Public Health. 2022 Jul;17(7):1113-1135. doi: 10.1080/17441692.2021.1919734. Epub 2021 May 2. PMID 33938368
- [Result] PREVAIL III Study Group; Sneller MC, Reilly C, Badio M, Bishop RJ, Eghrari AO, Moses SJ, Johnson KL, Gayedyu-Dennis D, Hensley LE, Higgs ES, Nath A, Tuznik K, Varughese J, Jensen KS, Dighero-Kemp B, Neaton JD, Lane HC, Fallah MP. A Longitudinal Study of Ebola Sequelae in Liberia. N Engl J Med. 2019 Mar 7;380(10):924-934. doi: 10.1056/NEJMoa1805435. PMID 30855742